CLINICAL TRIAL: NCT07077928
Title: Effects of Upgrading From Right Ventricular Pacing to Cardiac Resynchronization Therapy and Comparison With Dual-Chamber Defibrillator
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Professor Doctor, Bursa Postgraduate Hospital
Other Study IDs: Bursa PH CRT Upgrade
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Ventricular Arrhythmias and Cardiac Arrest
Keywords: Heart failure; Cardiac Resynchronization Therapy; Upgrade; Defibrillator; Pacemaker
MeSH Terms: conditions — Heart Failure; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pacemaker upgrade — CRT upgrade

SUMMARY:
Patients who consecutively underwent de novo CRT implantation, CRT upgrade, and DDDR ICD implantation at the Cardiology Clinic of Bursa Postgraduate Hospital between January 2019 and December 2023 according to the European Society of Cardiology (ESC) guideline criteria were included in the study.

DETAILED DESCRIPTION:
100 patients receiving de-novo CRT, 38 patients upgrading from RV pacing to CRT, and 169 patients receiving a DDDR-ICD implantation were included the study. Inclusion criteria were left ventricular ejection fraction lower than 35% and either QRS longer than 130ms for CRT groups or QRS≤120ms for the DDDR-ICD group. Primary endpoints were all-cause mortality and hospitalization for heart failure during a follow-up period extending up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

De novo CRT group:

* Sinus rhythm,
* age higher than 18,
* EF lower than 35%,
* New York Heart Association (NYHA) class II-IV,
* QRS >130 ms,
* patients with atrial fibrillation (AF) who converted to sinus rhythm and who remained symptomatic despite 3-6 months of guideline-directed medical therapy.

CRT upgrade group:

* Sinus rhythm,
* age higher than 18,
* EF lower than 35%,
* NYHA class II-IV,
* QRS duration >130 ms with RV pacing,

  -> 20% RV pacing rate,
* patients with AF who converted to sinus rhythm, at least 6 months since pacemaker implantation, and symptomatic despite 3-6 months of guideline directed medical therapy.

DDDR ICD group:

* Sinus rhythm,
* age higher than 18,
* EF lower than 35%,
* QRS ≤120 ms,
* NYHA class II-IV,
* patients with AF converted to sinus rhythm,
* receiving guideline-directed medical therapy.

Exclusion Criteria:

* patients with atrial fibrillation
* LV EF higher than 50 %
* NYHA Class 1
* Patients with active infection or cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who consecutively underwent de novo CRT implantation, CRT upgrade, and DDDR ICD implantation at the Cardiology Clinic Heart failure group in Sinus rhythm
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
All cause mortality and hospitalization for heart failure | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Hastanesi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No